CLINICAL TRIAL: NCT07158320
Title: Relaxation Training for Vasomotor Symptoms and Body Awareness in Menopausal and Postmenopausal Women
Brief Title: Relaxation Training for Menopausal and Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, PT,PHD,Prof., Baskent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KA 21/293
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Menopausal and Postmenopausal Women
Keywords: Menopause; Women's Health; Relaxation Therapy
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menopausal period group (Experimental): 24 individuals in the menopausal period
  Interventions: Behavioral: Relaxation training
- Postmenopausal period group (Experimental): 24 individuals in the postmenopausal period (patients who have been without a menstrual period for 12 months)
  Interventions: Behavioral: Relaxation training

INTERVENTIONS:
Behavioral: Relaxation training — In Jacobson's progressive muscle relaxation method, the first step is to make various muscle groups contract, to realize what it feels like to contract in this body area; The second step is to release these contracted muscle groups and notice how a relaxed muscle feels as the contraction subsides. During the exercise, the contraction is continued for 5 seconds. After the contraction, the muscles are relaxed for 10-15 seconds and in the meantime, rest is provided. Before starting the training, the person is taught the correct breathing technique and is asked to use the correct breathing technique throughout the practice. The practice should be done calmly without haste. During the practice, people should choose clothes that they can feel comfortable in. The practice should be applied in a quiet, dim environment where people can feel comfortable. It can also be performed with the eyes closed.

SUMMARY:
Relaxation training is one of the methods used in the reduction of many menopausal symptoms such as vasomotor symptoms, sleep disturbance, and emotional status changes.

Symptoms seen during menopause; sleep disturbance and lack of body awareness negatively affect women's daily lives. Relaxation exercises play an important role for women to manage this process better. In previous studies, the effects of relaxation training on hot flashes have been investigated, but a comprehensive study including body awareness and sleep problems has not been conducted yet. The aim of this study is to investigate the effect of relaxation training on vasomotor symptoms and body awareness in menopausal and postmenopausal periods.

ELIGIBILITY:
Inclusion Criteria:

* Being between 50-65 years old,
* Going through menopause period naturally
* People who do not receive hormone therapy

Exclusion Criteria:

* Who entered menopause surgically or medically,
* With a history of cancer,
* Who take hormone therapy,
* With neurological disease,
* Who use anti-symptom medication.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — menopausal and postmenopausal women
Enrollment: 48 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Menopausal symptoms evaluation scale (MSRS) | 6 weeks
  MSRS was developed by Schneider et al (2000) to measure the severity of general menopausal symptoms. The scale consists of 11 items in total and each item is scored between 0 and 4. Scoring was graded as 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. The highest score on the scale is 44, and the lowest score is 0. The increase in the scale score indicates the increase in the severity of the complaint.
Pittsburhg sleep quality scale (PSQS) | 6 weeks
  PSQS is an index that evaluates sleep problems and sleep quality in the last month, consisting of a total of 7 sub-components and 18 problems. These components are subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), use of sleeping pills (component 6) and daytime dysfunction (component 7). Each component is evaluated with a minimum of 0 and a maximum of 3 points. The scale total score is 0 at the lowest and 21 at the highest. According to the scale scoring, a score of 5 and above indicates that sleep quality is low.
Body awareness questionnaire | 6 weeks
  The body awareness questionnaire is a questionnaire consisting of four subgroups (changes in body process, sleep-wake cycle, estimation at the onset of the disease, estimation of body responses) aiming to determine the normal or abnormal sensitivity level of body composition. It includes 18 questions that measure various aspects of body consciousness, such as the ability to recognize physical sensations, engagement with the body, and awareness of physical condition in different circumstances. Each item is evaluated with a minimum of 1 and a maximum of 7 points. A high score indicates a high level of body awareness.
Body perception scale | 6 weeks
  Body perception scale is a scale that determines the satisfaction of the person with 40 different body parts or functions. The scale consists of 40 items and each item is scored between 1 and 5 (1 = I like it very much, 2 = I like it a lot, 3 = I am undecided, 4 = I do not like it very much; 5 = I do not like it at all). The total scale score is between 40 and 200. A high scale score indicates a decrease in satisfaction, and a low score indicates an increase in satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Ozunlu Pekyavas, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided